CLINICAL TRIAL: NCT00330811
Title: B-type Natriuretic Peptide in the Non-Cardiac Pediatric Patient
Status: Completed | Type: Observational
Sponsor: Emory University (Other)
Responsible Party: Principal Investigator, Kevin O. Maher, MD, Associate Professor of Pediatrics, Emory University
Other Study IDs: 1409-2005
Record Dates: First submitted 2006-05-25; First posted 2006-05-29 (Estimated); Last update posted 2016-12-02 (Estimated); Status verified 2016-11

CONDITIONS: Heart Diseases
Keywords: Pediatrics; Non-cardiac Illness; B-type Natriuretic Peptide (BNP)
MeSH Terms: conditions — Heart Diseases

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
B-type Natriuretic Peptide (BNP) is a hormone that is made by the pumping chambers of the heart. The BNP level can be measured by a blood test and is used as a marker for heart problems in adults. Deciding if a child has a heart problem or a lung problem can be very difficult, especially in infants. Several studies have demonstrated that BNP levels are elevated when children have heart disease.

The overall goal of the study is to be able to prove that obtaining BNP levels in pediatric patients can be used to identify heart problems. We already know that kids with heart problems have high BNP levels (>200pg/ml). We need to prove that children who come to the Emergency Department for non-cardiac problems still have normal BNP levels (<100pg/ml, slightly higher in the newborn population). This will be done by comparing BNP levels with the final diagnosis made by the ED physician.

DETAILED DESCRIPTION:
Introduction At Children's Healthcare of Atlanta, thousands of children are seen in the Emergency Department (ED) each year for evaluation and treatment. Deciding if a child has a cardiac or pulmonary problem can be very difficult, especially in infants. Early recognition of cardiac disease can significantly impact the physician's ability to provide appropriate treatment, make necessary interventions, and affect patient outcome. An accurate laboratory marker of cardiac disease for pediatric Emergency Medicine does not exist. B-Type Natriuretic Peptide (BNP) is a hormone produced by the ventricular myocardium (heart muscle) in response to increased myocardial demands. It has been used extensively in the adult population to evaluate patients for heart disease, and has been demonstrated to be very accurate in the differentiation of heart disease from lung disease in the adult Emergency Department.

There is increasing experience with BNP in pediatrics for the evaluation of heart disease, primarily in patients with congenital heart disease. The normal BNP level is less than 100 pg/ml, slightly higher in neonates. Patients who present to the ED and are diagnosed with heart disease are often admitted to the Cardiac Intensive Care Unit (CICU) for further management and stabilization. Part of the initial evaluation is a BNP level. These patients usually have marked elevation of the BNP levels in the 2000-5000 pg/ml range upon admission. The level varies with the type and severity of their heart disease. However very little is known about the non-cardiac ED patient BNP level. To utilize BNP as an accurate marker of cardiac disease in the pediatric ED, a clear difference between cardiac and non-cardiac patients needs to be demonstrated. If a large difference in BNP levels exists for the pediatric patient with heart disease who presents to the ED when compared to the child who presents to the ED with other non-cardiac disease processes, a useful marker of heart disease in children would be demonstrated.

Objectives: The objective of the proposed research is to determine the typical BNP level in non-cardiac pediatric patients who present to the ED for evaluation of respiratory and/ or infectious processes. The endpoint of the project will be the collection of BNP levels from 100 patients less than 6 years of age.

Hypothesis 1 (H1): BNP levels for children with non-cardiac disease will be in the normal range (< 100pg/ml), and can be easily distinguished from the elevated levels seen in children with congenital or acquired heart disease.

ELIGIBILITY:
Inclusion Criteria:

* Any child presenting to the pediatric ED at Children's Healthcare of Atlanta (CHOA)at Egleston undergoing evaluation for respiratory and/or infectious disease.
* Patient age is less than 6 years old.
* Patients having venipuncture for lab studies as a part of the ED admission.
* Informed consent being obtained from the legal guardians.

Exclusion Criteria:

* Patients with known congenital or acquired heart disease.
* Patients with previously diagnosed systemic disease such as malignancy, HIV, cystic fibrosis, organ transplant recipients.
* Patients that will not be having venipuncture for lab studies as a part of the ED admission.
* Trauma patients or those presenting with broken bones, dog bites, etc. (non-infectious presentation.)

Ages: 1 Day to 5 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Any child who is less than 6 years old seen in the Emergency Department evaluated for respiratory and/or infectious disease with order/s to have blood draw.
Sampling Method: Non-Probability Sample
Enrollment: 87 (Actual)
Dates: Start 2006-04; Primary Completion 2007-01 (Actual); Study Completion 2007-05 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kevin O Maher, MD, Principal Investigator — Emory University
Locations (1):
- Children's Healthcare of Atlanta, Atlanta, Georgia, United States